CLINICAL TRIAL: NCT00849407
Title: Genetic Risk Factors and Acquired Oncogenic Mutations of Melanoma
Acronym: M3
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Ichiro Okamoto, associate professor, Medical University of Vienna
Other Study IDs: M3-I
Record Dates: First submitted 2009-02-20; First posted 2009-02-23 (Estimated); Last update posted 2019-03-07 (Actual); Status verified 2019-03

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: melanoma patients
- 2: controls

SUMMARY:
Though it is generally accepted that exposure to sunlight is a major causative factor for skin cancer, the risk for developing melanoma is not directly linked to sun exposure such as in non-melanoma skin cancer. Therefore, a dual pathway has been proposed, distinguishing melanoma that develops on skin that is chronically exposed to sunlight from those that occur on skin that is normally protected. The risk for each type of melanoma is believed to be determined in part by genetic factors. To define these markers reproducibly, the investigators plan to establish a large cohort with comprehensive information regarding sun sensitivity (skin type), history of experienced sun exposure, skin pigmentation phenotypes, total number of nevi, and other types of skin tumors in a central European population. The investigators will obtain blood from all participants for DNA as well as serum analyses. Based on the finding that genetic variants of the melanocortin-1 receptor (MC1R) gene, associated with red hair and fair skin, have been shown to be associated with increased risk for melanoma, particularly those harboring BRAF mutations, the investigators will now focus on the study of recently discovered genetic variants associated with pigmentation. Furthermore, the investigators will study the relation of these variants with oncogenic mutations of melanoma in BRAF, RAS and c-Kit. The study of other genetic variants will follow, once a sufficiently large cohort has been established to reveal an independent genetic risk factor in a multivariate analysis including potential covariates as mentioned above. The identification of genetic risk factors for melanoma will not only help identify individuals with increased risk but also improve our understanding of the molecular background of the development of melanoma.

ELIGIBILITY:
Inclusion Criteria:

* patients with or without melanoma

Exclusion Criteria:

* HIV and Hepatitis C positive individuals.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Our goal is to recruit at least one thousand melanoma patients of any stage and one thousand controls in order to acquire a well sized cohort for identifying independent molecular markers in multivariate analyses (for statistical considerations see "Statistical analysis" on page 8). Patients who visit the out-door clinic of the Department of Dermatology at the Medical University of Vienna with any other diseases than melanoma, their spouses and spouses of melanoma patients will be asked to contribute as controls.
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2008-10; Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
melanoma | 2 years

SECONDARY OUTCOMES:
survival | 10 years

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Vienna, Austria